CLINICAL TRIAL: NCT03732131
Title: Long Term Safety and Efficacy of Faecal Microbiota Transplantation: a Nationwide Obeservational Study
Brief Title: The Finnish Faecal Microbiota Transplantation Study (FINFMT)
Acronym: FINFMT
Status: Recruiting | Type: Observational
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: University of Helsinki (Other); Helsinki University Central Hospital (Other); Turku University Hospital (Other Government); Tampere University Hospital (Other); Oulu University Hospital (Other); Kuopio University Hospital (Other); South Karelia, Social and Health Care District (Other); North Karelia Central Hospital (Other); Keski-Pohjanmaa Central Hospital (Unknown); Seinajoki Central Hospital (Other); Jyväskylä Central Hospital (Other); Kanta-Häme Central Hospital (Other Government); Mikkeli Central Hospital (Other); Vaasa Central Hospital, Vaasa, Finland (Other); Lapland Central Hospital (Unknown); Satakunta Central Hospital (Other); Kymenlaakso Social and Health Services (Unknown); Kainuu Social and Health Care Joint Authority (Other)
Responsible Party: Sponsor
Other Study IDs: HUS/3198/2017
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Faecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study is to follow up the long term effects of faecal microbiota tranplantation (FMT). All the over 18 years old patients receiving FMT and not included in other trials meet inclusion criteria to this study. Patients will be asked for a written consent. The outcome and possible side effects of the FMT will be followed by blood and feces samples for one year and with questionaires up to ten years after the FMT.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years age
* receiving FMT for rCDI or any other madical condition
* written consent
* Not included in other FMT trials

Exclusion Criteria:

* Unable to provide written consent
* < 18 years age
* Included in other FMT-trial

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Finnish patients over 18 years of age. Receiving FMT for recurring Clostridium difficile infektion (rCDI) which is the only indication for FMT. If experimental FMT would be given for any other condition after a throughout work up of a collegue of experts such a patien would meet inclusion criteria as well.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
The long term effects of FMT -questionnaire | 10 years
  The questionnaire has 52 questions. Weight and height are asked and appearance of certain symptoms. The answers are mostly yes or no. The questionnaire is not validated and it is descriptive and the answers are not scored.

CONTACTS AND LOCATIONS:
Overall Officials: Perttu Arkkila, PhD, Study Director — Head of Department
Locations (1):
- Joint Authority for Päijät-Häme Social and Health Care, Lahti, Finland

IPD SHARING:
Plan to Share IPD: No